CLINICAL TRIAL: NCT04787159
Title: Endometrial Cancer, a New Prospective Towards an Individually Adjusted Management Plans: A Multicenter International Study
Brief Title: Endometrial Cancer International Database
Acronym: ECID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: Middle-East OBGYN Graduate Education Foundation (Other)
Responsible Party: Principal Investigator, Sherif Abdelkarim Mohammed Shazly, Assistant lecturer, Assiut University
Other Study IDs: EC-ID21
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Endometrial Cancer
Keywords: carcinoma of corpus uteri; uterine malignancy; FIGO staging; adenocarcinoma; lymphadenectomy; hystrectomy; prognosis; prediction; machine learning
MeSH Terms: conditions — Endometrial Neoplasms; Adenocarcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project aims to determining prognostic factors and individualizing management decision per patient characteristics and endometrial cancer features. This study will include at least 10 centers from different countries that present at least Europe, South America, Asia, and Africa. Data will be retrospectively collected from January 2008 to December 2015 with a total follow-up of at least 5 years (December 2020).

DETAILED DESCRIPTION:
Endometrial cancer (EC) or carcinoma of corpus uteri is a neoplastic change, mostly adenocarcinoma, arising from uterine columnar epithelial lining. Abnormal uterine bleeding is the main presenting symptom especially in postmenopausal women. EC is estimated to be the seventh most commonly diagnosed cancer in women. It is considered the 16th leading cause of death in women with cancer worldwide, with 382 000 estimated new cases and 89 900 deaths in 2018. Factors as obesity, parity, diabetes mellitus, unopposed estrogen exposure, genetics and hormonal therapies are recognizable risks for EC. Other factors as chronic comorbidities, tumor size and organ metastasis influence staging, prognosis, and management protocols.

FIGO staging has been adopted as the standard classification system in the management of endometrial cancer. However, this staging system does not consider all factors that affect treatment decision and prognosis including but not limited to patient demographics, tumor grade, and lymphovascular space invasion. In addition, some interventions are still debatable particularly in the presence of intermediate disease e.g, grade II early EC. Available evidence supports combined pelvic and para-aortic lymphadenectomy in management of patients with EC. However, combined pelvic and para-aortic lymphadenectomy carry the risk of long term morbidities as lymphedema. Thus, hysterectomy alone as management plan is suggested in patients with low risk EC. More comprehensive studies of the multiple confounders that determine patient's risk are essential to reach an individually adjusted management plans and to predict prognosis of each individual case. Therefore, availability of large multicenter studies will provide robust evidence regarding optimal management of EC and hence, improve treatment outcome and prognosis particularly in the era of machine learning and artificial intelligence.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with endometrial cancer, between 2008 and 2015.
* Women should be diagnosed and managed by the corresponding center.
* Patients with adequate clinical and pathological data.

Exclusion Criteria:

* Inadequate information and follow-up for at least 5 years.
* Authorization to use anonymous patient data for research purposes.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All women who were diagnosed with endometrial cancer at any stage, of all histological types and grades, between 2008 and 2015.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival at 1 year | At 1 year
  Number of women who are alive after cancer treatment divided by total number of patients at study onset
Overall survival at 3 years | At 3 years
  Number of women who are alive after cancer treatment divided by total number of patients at study onset
Overall survival at 5 years | At 5 years
  Number of women who are alive after cancer treatment divided by total number of patients at study onset
disease free survival at 1 year | At 1 year
  Number of women who are are disease free after cancer treatment divided by total number of patients at study onset
disease free survival at 3 years | At 3 years
  Number of women who are are disease free after cancer treatment divided by total number of patients at study onset
disease free survival at 5 years | At 5 years
  Number of women who are are disease free after cancer treatment divided by total number of patients at study onset

CONTACTS AND LOCATIONS:
Overall Officials: Sherif A Shazly, M.Sc, Principal Investigator — Assiut University

REFERENCES:
- [Background] Bell DW, Ellenson LH. Molecular Genetics of Endometrial Carcinoma. Annu Rev Pathol. 2019 Jan 24;14:339-367. doi: 10.1146/annurev-pathol-020117-043609. Epub 2018 Oct 17. PMID 30332563
- [Background] Lax SF. [New features in the 2014 WHO classification of uterine neoplasms]. Pathologe. 2016 Nov;37(6):500-511. doi: 10.1007/s00292-016-0230-4. German. PMID 27738815
- [Background] Hamilton CA, Pothuri B, Arend RC, Backes FJ, Gehrig PA, Soliman PT, Thompson JS, Urban RR, Burke WM. Endometrial cancer: A society of gynecologic oncology evidence-based review and recommendations, part II. Gynecol Oncol. 2021 Mar;160(3):827-834. doi: 10.1016/j.ygyno.2020.12.024. Epub 2021 Jan 13. PMID 33451724
- [Background] Soja M, Masternak M, Piwowarczyk I, Janas L, Szyllo K, Nowak M. Analysis of the results of invasive diagnostic procedures in patients referred to gynecologic department due to abnormal uterine bleeding. Prz Menopauzalny. 2020 Dec;19(4):155-159. doi: 10.5114/pm.2020.101942. Epub 2021 Jan 7. PMID 33488325
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Ignatov A, Ortmann O. Endocrine Risk Factors of Endometrial Cancer: Polycystic Ovary Syndrome, Oral Contraceptives, Infertility, Tamoxifen. Cancers (Basel). 2020 Jul 2;12(7):1766. doi: 10.3390/cancers12071766. PMID 32630728
- [Background] Raglan O, Kalliala I, Markozannes G, Cividini S, Gunter MJ, Nautiyal J, Gabra H, Paraskevaidis E, Martin-Hirsch P, Tsilidis KK, Kyrgiou M. Risk factors for endometrial cancer: An umbrella review of the literature. Int J Cancer. 2019 Oct 1;145(7):1719-1730. doi: 10.1002/ijc.31961. Epub 2019 Feb 20. PMID 30387875
- [Background] Kruse AJ, Ter Brugge HG, de Haan HH, Van Eyndhoven HW, Nijman HW. Vaginal hysterectomy with or without bilateral salpingo-oophorectomy may be an alternative treatment for endometrial cancer patients with medical co-morbidities precluding standard surgical procedures: a systematic review. Int J Gynecol Cancer. 2019 Feb;29(2):299-304. doi: 10.1136/ijgc-2018-000015. Epub 2019 Jan 18. PMID 30659027
- [Background] Murali R, Delair DF, Bean SM, Abu-Rustum NR, Soslow RA. Evolving Roles of Histologic Evaluation and Molecular/Genomic Profiling in the Management of Endometrial Cancer. J Natl Compr Canc Netw. 2018 Feb;16(2):201-209. doi: 10.6004/jnccn.2017.7066. PMID 29439179
- [Background] Petousis S, Christidis P, Margioula-Siarkou C, Papanikolaou A, Dinas K, Mavromatidis G, Guyon F, Rodolakis A, Vergote I, Kalogiannidis I. Combined pelvic and para-aortic is superior to only pelvic lymphadenectomy in intermediate and high-risk endometrial cancer: a systematic review and meta-analysis. Arch Gynecol Obstet. 2020 Jul;302(1):249-263. doi: 10.1007/s00404-020-05587-2. Epub 2020 May 28. PMID 32468162
- [Background] Mariani A, Webb MJ, Keeney GL, Haddock MG, Calori G, Podratz KC. Low-risk corpus cancer: is lymphadenectomy or radiotherapy necessary? Am J Obstet Gynecol. 2000 Jun;182(6):1506-19. doi: 10.1067/mob.2000.107335. PMID 10871473
- [Background] Reijnen C, Gogou E, Visser NCM, Engerud H, Ramjith J, van der Putten LJM, van de Vijver K, Santacana M, Bronsert P, Bulten J, Hirschfeld M, Colas E, Gil-Moreno A, Reques A, Mancebo G, Krakstad C, Trovik J, Haldorsen IS, Huvila J, Koskas M, Weinberger V, Bednarikova M, Hausnerova J, van der Wurff AAM, Matias-Guiu X, Amant F; ENITEC Consortium; Massuger LFAG, Snijders MPLM, Kusters-Vandevelde HVN, Lucas PJF, Pijnenborg JMA. Preoperative risk stratification in endometrial cancer (ENDORISK) by a Bayesian network model: A development and validation study. PLoS Med. 2020 May 15;17(5):e1003111. doi: 10.1371/journal.pmed.1003111. eCollection 2020 May. PMID 32413043